CLINICAL TRIAL: NCT00622791
Title: Effects of Cardiopulmonary Bypass on Plasma Propofol Concentrations and Bis Values During Coronary Surgery
Brief Title: Propofol Pharmacokinetics and Pharmacodynamics During Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Maria J. C. Carmona, Faculdade de Medicina da Universidade de São Paulo
Other Study IDs: 802-01
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2008-02-25 (Estimated); Status verified 2008-02

CONDITIONS: Coronary Artery Disease; Cardiopulmonary Bypass; Coronary Artery Bypass Graft
Keywords: Cardiopulmonary bypass; coronary artery bypass graft; coronary artery disease; propofol; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CABG group: Patients undergoing coronary artery bypass graft with cardiopulmonary bypass
- OPCAB group: Patients undergoing off-pump coronary artery bypass graft

SUMMARY:
Cardiopulmonary bypass (CPB) is known to alter pharmacokinetics (PK) and brain sensitivity to several drugs, including propofol. Few studies, however, have tested if propofol pharmacokinetical alterations observed after CPB could contribute to the increased hypnotic effect of propofol after CPB. This study was designed to test the hypothesis that changes in the PK of propofol contribute to an increase in its hypnotic effects after CPB as evidenced by changes in bispectral index (BIS) values.

Twenty undergoing coronary artery bypass graft patients will be allocated in two groups: 1) CPB groups and 2) off-pump coronary artery bypass graft. Bispectral Index values and blood samples for plasma propofol concentration measurements will be collected along the surgery and up to 12 hours in the post-operative period. Plasma propofol concentrations, Bispectral index values and propofol PK will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Isolated coronary artery bypass indication
* Left ventricular ejection fraction greater than 50 %
* Absence of preoperative pulmonary dysfunction

Exclusion Criteria:

* Intra and postoperative circulatory shock
* Postoperative pulmonary dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty patients undergoing elective coronary artery bypass graft surgery
Sampling Method: Probability Sample
Enrollment: 20 (Actual)

PRIMARY OUTCOMES:
Propofol pharmacodynamics and pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Maria M Carmona, MD PhD, Principal Investigator — Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Barbosa RA, Santos SR, White PF, Pereira VA, Silva Filho CR, Malbouisson LM, Carmona MJ. Effects of cardiopulmonary bypass on propofol pharmacokinetics and bispectral index during coronary surgery. Clinics (Sao Paulo). 2009;64(3):215-21. doi: 10.1590/s1807-59322009000300012. PMID 19330248